CLINICAL TRIAL: NCT01324882
Title: Study to Examine Insertion of 2 Colonoscopes Trial
Brief Title: Colonoscope Insertion Trial Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Joseph Anderson, Associate Prof (Adjunct), UConn Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 10-246-1; 1-642-01 (Other: UCHC)
Record Dates: First submitted 2011-03-24; First posted 2011-03-29 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Colorectal Cancer
Keywords: colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Arm (Experimental): This is the group who will have a colonoscopy with the Olympus Technically Improved Colonoscope.
  Interventions: Device: Colonoscopy with Olympus Technically Improved Colonoscope
- Control (Active Comparator): This is the group who will have a colonoscopy with the traditional colonoscope Olympus CF-H180.
  Interventions: Device: Control with standard colonoscope Olympus CF-H180

INTERVENTIONS:
Device: Colonoscopy with Olympus Technically Improved Colonoscope — The standard colonoscopy will be performed using the Olympus Technically Improved Colonoscope.
  Other Names: Olympus Technically improved colonoscope
  Arms: Study Arm
Device: Control with standard colonoscope Olympus CF-H180 — Standard colonoscopy using the adult scope, Olympus CF-H180.
  Other Names: Olympus CF-H180
  Arms: Control

SUMMARY:
This research study is about determining how well a Technically Improved Colonoscope from Olympus works in helping the doctor in guiding the scope through the large bowel or colon. When a doctor performs a colonoscopy he guides or inserts the scope from the rectum to the appendix where the small bowel ends and the large bowel begins. There are points during this insertion where there are turns in the colon which can create a loop in the colonoscope. These loops can stretch the colon and create some discomfort and also require special maneuvers by the nurse or patient to help reduce or minimize the loop. Thus, reducing the looping will make it more comfortable for the patient and more efficient for screening for polyps. The purpose of the study is to examine this colonoscope and compare it to the traditional adult colonoscope (Olympus CF-H180). The investigators hypothesis is that this colonoscope will function better with regard to insertion of the scope from the rectum to the cecum.

DETAILED DESCRIPTION:
There will be two arms to the study, the CF-H180 adult colonoscope (Control Arm) and the Olympus Technically Improved Colonoscope (Olympus). (Control Arm). In this protocol the investigators will randomize patients to either the adult colonoscope or to the Olympus Technically Improved Colonoscope (Olympus) arm. The name of the arm (CF-H180 adult colonoscope or Technically Improved Colonoscope) will be in a sealed envelope and opened by the nurse. The endoscopist will be blinded to the scope that will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for outpatient colonoscopy between the ages of 35 and 75 years of age
* The patient population will be open. However, it is known that thin female patients (BMI < 25) and/or past history of diverticular disease and/or gynecological surgery and men & women who are tall (6'+) and patients with constipation are usually difficult candidates for a complete colonoscopy (retroflex in the cecum)
* Adequate bowel preparation
* The ability to provide informed consent

Exclusion Criteria:

* Women that are pregnant
* Patients with a past history of inflammatory bowel disease
* Patients with a past history of surgical resection (hemicolectomies, etc)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C Anderson, M.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from study initiation 1/31/2011 until June 30,2011. Patients were recruited from the clinic.
Pre-assignment Details: No details to report
Period: Overall Study
Arm/Group | Study Arm | Control
Started | 27 (27 patients were randomized to this arm.) | 30 (30 patients were randomized to this arm)
Completed | 27 (27 patients had the colonoscopy) | 30 (30 patients had the colonoscopy)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Arm | Control | Total
Number analyzed (Participants) | 27 | 30 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (6.8) | 56 (8.3) | 55.85 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  United States | 27 | 30 | 57

OUTCOME MEASURES:

1. Primary Outcome: Time to Intubate the Cecum
Description: The time in seconds that it required to intubate the cecum as defined in our protocol.
Time Frame: The outcome was measured during the colonoscopy which was Day 1. The duration of the study was the colonoscopy on Day 1. Once the colonoscopy was finished, the study was over.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Study Arm | Control
Number analyzed (Participants) | 27 | 30
seconds | 271 (196) | 403 (148)

2. Primary Outcome: Intubation of Cecum
Description: The ability of endoscopist to intubate the cecum with enough control of the tip to abut the appendix or begin to retroflex in the cecum.
Time Frame: (day 1) Within time for performance of colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm | Control
Number analyzed (Participants) | 27 | 30
Participants | 27 | 29
Statistical Analysis 1: Comparison: Study Arm vs Control; Test type: Other; p = 1.00, Fisher Exact

ADVERSE EVENTS:
Time Frame: An Average of 20 minutes, up to 30 minutes post procedure.
Arm/Group | Study Arm | Control
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/30
Other Adverse Events (participants affected / at risk) | 0/27 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No